CLINICAL TRIAL: NCT01970774
Title: Assessing Feasibility and Utility of Enhancing Medication Therapy Management With Pharmacist-Delivered Pharmacogenetic Testing
Brief Title: Medication Therapy Management With Pharmacogenetic Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00048123
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2014-10

CONDITIONS: Pharmacogenetics; Medication Therapy Management
MeSH Terms: interventions — myotubularin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MTM and PGx (Experimental): Participants attend two MTM sessions and have PGx testing
  Interventions: Other: MTM with PGx

INTERVENTIONS:
Other: MTM with PGx — Patients will attend MTM sessions and receive PGx testing

SUMMARY:
This study aims to investigate the benefit and feasibility of providing pharmacogenetic (PGx) testing as part of a standard medication therapy management (MTM) session for patients taking multiple medications, a high-risk population for adverse drug reactions and non-response. Research participants will attend two MTM sessions and undergo PGx testing to inform the MTM plan. Participants will also complete 2 surveys pre and post-MTM/PGx testing. Data analysis will assess the impact of MTM/PGx testing on recommendations for drug dosing, clinical outcomes, patient satisfaction, and feasibility of service delivery. Safety issues are minimal with the primary risks being associated with loss of confidentiality, typical discomfort associated with acquiring blood samples, and genetic discrimination.

ELIGIBILITY:
Inclusion Criteria:

* currently prescribed 3 medications, one of which must be simvastatin or clopidogrel
* 18 years of age or older
* English speaking
* patients of Mahesh Patel or William Kraus at Duke Southpoint Clinic

Exclusion Criteria:

* if patient has ever had MTM or PGx

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with MTM and PGx | 3 months after completion of MTM2
  This will be assessed by a quantitative survey
Change in clinical biomarkers associated with drug therapy | baseline and 2 months
  Changes in biomarkers before and after MTM/PGx will be measured. Biomarkers of study group will be compared to chart-review control
Number of recommended drug selection/dosing adjustments | approximately 9 months
  Drug selection/doing changes will be compared between study population and chart-review controls

SECONDARY OUTCOMES:
Physician time to perform MTM and PGx | end of study, approx. 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Haga, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Health Center at Southpoint, Durham, North Carolina, United States